CLINICAL TRIAL: NCT02509520
Title: Rehabilitation, NMES and High Protein to Reduce Post ICU Syndrome in the Elderly
Brief Title: Assessing The Effects of Exercise, Protein, and Electric Stimulation On Intensive Care Unit Patients Outcomes
Acronym: ExPrEs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Avelino Verceles, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00056749
Record Dates: First submitted 2015-07-21; First posted 2015-07-28 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Muscle Weakness; Critical Illness; Sarcopenia
Keywords: Nutritional supplementation; Neuromuscular Electric Stimulation; ICU acquired weakness; Post ICU Syndrome; sarcopenia
MeSH Terms: conditions — Muscle Weakness; Critical Illness; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobility-based Physical Rehab (MPR) (No Intervention): ICU control group receiving only mobility based rehabilitation (MPR).
- MPR and Neuromuscular Stimulation and HPRO (Active Comparator): ICU group receiving mobility based rehabilitation and NMES and High protein supplementation.
  Interventions: Dietary Supplement: MPR and High Protein Supplement (HPRO) and Neuromuscular Electric Stimulation (NMES)

INTERVENTIONS:
Dietary Supplement: MPR and High Protein Supplement (HPRO) and Neuromuscular Electric Stimulation (NMES) — The MPR provides strength and cardiopulmonary endurance training, which consist of exercises to promote function movements. Intensity is based on patient's hemodynamic responses and subjective report using Modified Borg Dyspnea Scale. Intensity, duration, or type of activity will be modified each session to achieve a moderately intense physiologic response. The NMES protocol requires self-adhesive surface electrodes be placed on quadriceps muscles and lower leg bilaterally, twice daily. This protocol is based on prior NMES protocols used to stimulate muscle protein synthesis in older diabetic patients, preserve muscle mass in intensive care patients and increase strength in older adults after knee replacement. The HPRO intervention is based on caloric needs, calculated using validated equations to maintain positive nitrogen balance. Protein will be supplemented as isolated amino acids twice/day to deliver ~15g of essential amino acids per serving, with a goal of 1.6 g/kg/day.
  Arms: MPR and Neuromuscular Stimulation and HPRO

SUMMARY:
Elderly patients who experience a prolonged ICU stay are at high risk for developing post intensive care unit syndrome (PICS), a serious medical condition manifested by loss of muscle mass, weakness, malnutrition and neurocognitive decline. PICS often leads to chronic disability, prolonged mechanical ventilation and the need for costly extended stays in long term care facilities (LTCs). The investigators' preliminary study shows attempts at rehabilitating patients who have already developed PICS are minimally effective, resulting in only modest improvements in functionality. This project will determine the effects of mobility-based physical rehabilitation (MPR) combined with neuromuscular electric stimulation (NMES) and high protein supplementation (HPRO) early in a patients ICU stay on preventing PICS related musculoskeletal and functional deficits, and improving clinical outcomes.

DETAILED DESCRIPTION:
Older, critically ill patients who survive their ICU stay frequently develop post-ICU syndrome (PICS) - a condition manifested by sarcopenia, weakness, malnutrition and neurocognitive decline - which occurs as a result of a critical illness, prolonged bed rest, catabolism, and polypharmacy. PICS frequently leads to chronic disability, prolonged mechanical ventilation (MV), functional deficits, and the need for extended rehabilitation in long term care facilities (LTCs). As the majority of patients admitted to ICUs are ≥ 65 years old, many of these patients are at high risk for PICS. Since the care of ICU patients is primarily focused on the medical management of the acute critical illness, there are limited resources and strategies available to prevent PICS. Evidence suggests mobility-based physical rehabilitation (MPR) combined with resistive training with neuromuscular electric stimulation (NMES) and high protein diets (HPRO) containing essential amino acids can mitigate the loss of muscle mass and function during bed rest in the elderly. The investigators hypothesize that preventive therapy involving the addition of both NMES and HPRO to MPR early and throughout the ICU and hospital stay can mitigate PICS-associated sarcopenia, malnutrition, and immobility to confer valuable health benefits toward recovery. To test this, the investigators will use a 2x2 factorial design in which older, MV ICU patients will all receive comprehensive ICU care and MPR, then be randomized to one of 4 groups: 1) MPR+NMES, 2) MPR+HPRO, 3) all 3 together, or 4) MPR alone (control), to determine independent and combined effects of the interventions.

The Specific Aims are to 1) determine the effects of adding NMES and HPRO interventions to MPR on muscle mass, strength, and mobility function in older, critically ill MV patients while still in the ICU, and 2) determine the effects of adding NMES and HPRO interventions to MPR on the clinical outcomes of time to weaning from MV, ICU/hospital length of stay and discharge disposition of these patients.

This proposal capitalizes on the interdisciplinary collaboration among Pulmonary/Critical Care Intensivists, Physical Therapists, Geriatricians, Clinical Nutritionists, Statisticians and Nutrition and Metabolism clinical researchers examining the efficacy of the proposed comprehensive rehabilitation approach. The investigators' primary goal is to attenuate the severity of sarcopenia and functional decline in this older, critically ill population at risk for severe disability. Additionally, by focusing on maintaining skeletal muscle mass, function, and strength, the investigators hope to improve clinical outcomes. The investigators posit this combined therapy will mitigate PICS-associated disability and speed the recovery from critical illness in older, MV ICU patients. This project has high overall impact as the intervention is easily administered by hospital staff and may greatly reduce the physiological and functional declines while hastening recovery during acute ICU hospitalization in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Respiratory insufficiency requiring mechanical ventilation (MV)
* ICU presentation < 6 days
* Patient or legally authorized representative able to provide written or witnessed verbal informed consent in English
* All four limbs intact and mobile
* Eligible for and able to participate in physical therapy
* Pre admission Barthel Index >70

Exclusion Criteria:

* Acute kidney injury with a glomerular filtration rate < 30 ml/min
* Diagnosis of severe organ dysfunction including end stage liver disease or cirrhosis
* Diagnosis of active cancer
* Acute or chronic organ transplant rejection
* Exceedingly high mechanical ventilator settings (FiO2>60%, PEEP>12) or alternative modes of mechanical ventilation (inverse ratio pressure control, airway pressure release ventilation)
* Severe functional impairment or physical impairment to rehabilitation
* On high dose vasopressor agents (> 5mcg of norepinephrine or equivalent)
* Liver function tests > 2.5 x normal limits (normal reference ranges include AST between 10 and 40 units/L or ALT between 7 and 56 units/L)
* Chronic dementia or cognitive impairment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 14 days
  Muscle mass as measured by lower extremity muscle volume
Global body strength | 14 days
  Muscle group strength as measured by hand held dynamometer and by hand grip strength
Mobility status | 14 days
  Outcome as measured by combined 6 minute walk distance and gait speed
Short Physical Performance Battery | 14 days
  Short Physical Performance battery will be assessed at baseline and at 7 and 14 days.

SECONDARY OUTCOMES:
Time to weaning | 14 days
  As measured by ventilator days
ICU/Hospital length of stay | 14 days
  Days in the ICU, days in the hospital
Discharge disposition | 30 days
  home, nursing home, acute rehabilitation, readmission, death, remains hospitalized
Weaning success | 14 days
  proportion of patient successfully weaned with in a 14 day period, and eventually

CONTACTS AND LOCATIONS:
Locations (1):
- U of Maryland, Baltimore, Professional Schools IRB, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verceles AC, Serra M, Davis D, Alon G, Wells CL, Parker E, Sorkin J, Bhatti W, Terrin ML. Combining exercise, protein supplementation and electric stimulation to mitigate muscle wasting and improve outcomes for survivors of critical illness-The ExPrES study. Heart Lung. 2023 Mar-Apr;58:229-235. doi: 10.1016/j.hrtlng.2022.11.013. Epub 2022 Dec 5. PMID 36473808